CLINICAL TRIAL: NCT00359060
Title: Physical Activity and Breast Cancer Risk in Postmenopausal Women: the SHAPE Study
Brief Title: Physical Activity and Breast Cancer Risk in Postmenopausal Women:the SHAPE Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government); Dutch Cancer Society (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UU 2003-2793
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-07

CONDITIONS: Breast Cancer
Keywords: Physical activity; Sex steroid hormones; Breast cancer risk; Intervention study; Postmenopausal women
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

INTERVENTIONS:
Behavioral: Physical activity

SUMMARY:
Purpose of the SHAPE study is to examine the effects of an 1-year exercise programme on endogenous hormone levels associated with breast cancer among sedentary postmenopausal women and whether a decrease in intra-abdominal fat is associated with a lowering of these hormone levels.

DETAILED DESCRIPTION:
Physical activity has been associated with a decreased risk for breast cancer. The biological mechanism(s) underlying the association between physical activity and breast cancer is not clear. Most prominent hypothesis is that physical activity may protect against breast cancer through reduced lifetime exposure to endogenous hormones. Another hypothesis is that physical activity prevents overweight and abdominal adiposity.

In this intervention study, 189 sedentary postmenopausal women who are aged 50-69 years are randomly allocated to an intervention or a control group. The intervention consists of an 1-year moderate-to-vigorous intensity aerobic and strength training exercise programme. Participants allocated to the control group are requested to retain their habitual exercise pattern. Primary study parameters measured at baseline, at four months and at 12 months are: serum concentrations of endogenous estrogens, endogenous androgens, sex hormone binding globulin and insulin. Other study parameters include: amount of total and abdominal fat, weight, BMI, body fat distribution, physical fitness, blood pressure and lifestyle factors.

This study will contribute to the body of evidence relating physical activity and breast cancer risk and will provide insight into possible mechanisms through which physical activity might be associated with reduced risk of breast cancer in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50 -69 year
* > 12 months since last menses
* Non-smokers (at least 12 months)
* Sedentary
* Knowledge of the Dutch language
* Agreement to be randomly assigned to either the exercise intervention or control group
* Informed consent to participate in all screening and study activities

Exclusion Criteria:

* Use of hormone replacement or oral contraceptives in past 6 months
* Morbidly obese (BMI > 40)
* BMI < 22
* Currently on or planning to go on a strict diet
* Ever diagnosed with breast cancer
* Diagnosis of other types of cancer in the past 5 years
* Diabetes mellitus or other endocrine related diseases
* Disorders or diseases (locomotor, optical, neurological, mental) that might impede the participation in the exercise programme
* Alcohol or drug abuse
* Maintenance use of corticosteroids
* Use of beta blockers

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2005-01; Study Completion 2006-09

PRIMARY OUTCOMES:
Serum concentrations of endogenous estrogens: estradiol (total, free), estrone, estrone sulfate
Serum concentrations of endogenous androgens: testosterone, androstenedione
Serum concentrations of sex hormone binding globulin
Serum concentrations of fasting insulin
Insulin sensitivity

SECONDARY OUTCOMES:
Amount of total body fat and intra-abdominal fat
Weight
Body Mass Index (BMI)
Body fat distribution
Waist to hip ratio
Physical Fitness
Blood pressure
Lifestyle parameters (covariates)
Exercise behaviour (habitual physical activity, past week activity, physical activity in the past)
Diet (daily caloric intake; percent daily calories from fat, carbohydrates and proteins)
Alcohol consumption
Medication use
Reproductive factors
Medical history

CONTACTS AND LOCATIONS:
Overall Officials: Jantine Schuit, PhD, Principal Investigator — Dutch Institute of Public Health and the Environment; Petra HM Peeters, PhD, Principal Investigator — University Medical Center Utrecht, Julius Center
Locations (1):
- University Medical Center Utrecht, Julius Center, Utrecht, Netherlands

REFERENCES:
- [Derived] Monninkhof EM, Peeters PH, Schuit AJ. Design of the sex hormones and physical exercise (SHAPE) study. BMC Public Health. 2007 Sep 4;7:232. doi: 10.1186/1471-2458-7-232. PMID 17767724